CLINICAL TRIAL: NCT02686515
Title: Comparative Effectiveness Research of Dual-task and Single-task Balance Training on Cognitive-motor Interference, Balance Confidence, Fall Prevention, Functional Performance, and Quality of Life in People With Stroke
Brief Title: Comparative Effectiveness Research of Dual-task and Single-task Balance Training in People With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Collaborators: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Li-Ling Chuang, Associated Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MOST104-2314-B-182-035-MY3
Record Dates: First submitted 2016-02-16; First posted 2016-02-19 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single-task balance training group (Active Comparator): Participants in the single-task training group will participate in 12-session programs administered for 60 minutes each session, 3 times per week for 4 weeks. They will start walking on a treadmill with a self-selected comfortable speed for 5 minutes of warm-up and then receive an individually-progressed program of balance training aimed at improving standing balance and walking abilities.
  Interventions: Device: single-task balance training
- Dual-task balance training group (Experimental): Participants in the dual-task training group will also participate in a 12-session program conducted 60 minutes per session, 3 days a week, for a total of 4 weeks. They will perform a cognitive task or motor task concurrently with the balance/gait task. The framework of progressive balance exercises in the dual-task training group will be progressed from simple to more complex tasks as outlined for the single-task training group. In addition, a variety of added tasks will be progressively integrated into the dual-task balance training program.
  Interventions: Device: dual-task balance training

INTERVENTIONS:
Device: single-task balance training — The framework of progressive balance exercises in the single-task training will include body stability tasks (Stance activities), transitional activities (Sit to stand and walk), and body transfer tasks (Gait activities). These exercises target various systems for balance control, such as stability limits (standing with changes in base of support and weight shifting), sensory orientation (standing on compliant surfaces with eyes open and eyes closed), postural responses (reactions to balance perturbation, sit to stand and walk), and gait (treadmill walking with increasing speed).
  Arms: Single-task balance training group
Device: dual-task balance training — Three cognitive tasks will be used for dual-task training while standing and walking: auditory discrimination tasks, verbal fluency tasks, and calculation tasks. In addition, motor tasks such as carrying a bag, holding a glass of water, alternating hand movement, carrying a tray with glasses, or getting keys out of a pocket will also be included as added tasks.
  Arms: Dual-task balance training group

SUMMARY:
The objective of this study is to investigate the effect of dual-task training at impairment, disability, and participation levels for stroke survivors and investigate possible factors affecting cognitive-motor interference (CMI) under dual-task conditions. Specifically, we will compare the immediate and retention effects of dual-task balance training and single-task balance training on CMI, balance confidence, fall rate, functional performance, and quality of life in individuals with stroke (Aim 1). The second aim of this study is to explore how lateralization, stroke chronicity, task type, and task difficulty may influence patterns of CMI (Aim 2). The third aim of this study is to investigate whether dual-task balance assessments are more sensitive than single-balance assessment in distinguishing stroke fallers from stroke non-fallers (Aim 3).

DETAILED DESCRIPTION:
Gait-related dual-task impairments are common problems experienced in people with stroke by walking more slowly or taking shorter steps in dual-task walking. Decrements in dual-task capacity may predispose stroke survivors to risk of falls and affect negatively on functional independence and quality of life. Currently there is a need to explore whether people with stroke practice dual-tasking in standing and walking will lead to enhance dual-task performance and reduce falls rate. However, there is a lack of prospective, controlled studies which quantify balance, gait, cognition, and fall-risk after dual-task training. The objective of this study is to investigate the effect of dual-task training at impairment, disability, and participation levels for stroke survivors and investigate possible factors affecting cognitive-motor interference (CMI) under dual-task conditions. Specifically, we will compare the immediate and retention effects of dual-task balance training and single-task balance training on CMI, balance confidence, fall rate, functional performance, and quality of life in individuals with stroke (Aim 1). The second aim of this study is to explore how lateralization, stroke chronicity, task type, and task difficulty may influence patterns of CMI (Aim 2). The third aim of this study is to investigate whether dual-task balance assessments are more sensitive than single-balance assessment in distinguishing stroke fallers from stroke non-fallers (Aim 3).

A prospective randomized control trial will be conducted at 2 medical centers in this study. Forty-eight people with stroke will be randomly allocated to either a single- or dual-task balance training group. Both groups will receive 12 hours of training over 4 weeks at progressively increasing task difficulty (60 minutes per session, three times a week, for four weeks). The single-task training group will undertake balance training and gait training. The dual-task training group will train the same set of balance activities as the single-task training while simultaneously performing a variety of added cognitive or motor tasks with instruction of a variable priority. During each session, participants in dual-task training practice shifting attention between tasks by spending half of the training attention focus on the balance task, and half focus on the secondary cognitive or motor task. A blinded assessor will conduct three assessments at baseline, post intervention, and 1-month follow-up. At baseline, all participants will be examine balance, gait, and cognitive performance under single-task (standing/walking at preferred speed and fast speed only, cognitive task only) and dual-task conditions (standing/walking at preferred speed and fast speed and concurrent cognitive task). Three cognitive tasks (simple auditory reaction time task, counting backward by 3s task, and Stroop task) will be used to examine patterns of CMI because these tasks represent different domains of cognitive function (information processing speed, working memory, and executive function). The primary outcome measure of cognition will be the composite score of accuracy and reaction time. The primary outcome measure of balance will be the sway index in mCTSIB test on a BioSway balance system under single- and dual-task standing. The primary outcome measure of gait will be gait speed on 10 m walk test under single- and dual-task walking. Secondary outcome measures will include: Berg Balance Scale, the Timed Up and Go test under single- and dual-task conditions, Activity-specific Balance Confidence Scale, Fugl-Meyer Assessment, Functional Independence Measure, Nottingham Extended Activities of Daily Living Scale, and Stroke Impact Scale. Additionally, falls will be prospectively monitored monthly and recorded during the following 6 months after the training. Repeated measure ANOVA will be used to compare measurements baseline, after training, and follow-up between the groups.

ELIGIBILITY:
Inclusion Criteria:

* first-ever stroke with onset duration more than 3 months
* able to walk with or without walking aids
* self-selected gait speed at least 0.6 m per second determined during a 10m walk test
* no severe vision, hearing, and language problems
* have experienced at least one fall in the previous year

Exclusion Criteria:

* have orthopedic condition affecting their gait or other diseases that might interfere with participation in the training program
* could not stand for at least two minutes without assistance
* score less than 24 on the Mini-Mental State Examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-03-02 (Actual); Primary Completion 2017-05-26 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Sway index | 10 minutes
  Participants will stand on a platform (Biosway Balance System, Biodex Medical Systems, Inc., NY, USA) and perform modified clinical test of sensory integration of balance test (mCTSIB) for 20 seconds in each of 4 conditions (Eyes open/closed, Firm/Foam surface). The instruction of this test is to maintain your center of balance and try not to move. The primary outcome of balance ability is sway index. The sway index is really the standard deviation of the sway angle. The higher the sway index the more unsteady the participant was during the test.
Gait speed | 5 minutes
  Participants will walk 10m at their preferred speed and at fast speed. Participants will be instructed to begin walking about 1 m before stepping on the walkway and to keep walking about 1 m beyond the walkway to exclude acceleration and deceleration phases on the walkway. The time to complete the middle 10 m will be recorded using a stopwatch. The primary outcome measure will be gait speed under single- and dual-task conditions.
Composite score = Accuracy/Reaction time | 10 minutes
  Participants will be asked to perform three different cognitive tasks while sitting, standing, walking at preferred speed, and walking at fast speed. The order of three cognitive tasks will be counterbalanced, but will be equal for the single- and dual-task conditions.These three cognitive tasks are simple reaction time task, counting backward by 3s, and Stroop task.To account for possible speed-accuracy trade-off, a composite score will be calculated by dividing accuracy (% correct responses) by verbal reaction time (milliseconds) will be used to indicate cognitive performance.
Cognitive-Motor Interference (CMI) | 30 minutes
  The effect of dual-tasking on both standing/walking and cognitive parameters will be assessed by comparing any change in performance of balance/gait and cognitive measures between single- and dual-task conditions. We will calculate CMI for each of the balance/gait outcome measures and 3 cognitive measures using following formula: [(Single-task - Dual-task)/Single-task *100]. Higher cost indicates poor performance on dual-task conditions.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | 5-10 minutes
  The BBS will be used to quantify balance performance under single-task conditions on tasks such as standing with eyes closed, standing with feet together, and picking up an object from the floor. Scores of the BBS range from 0 to 56, with higher scores suggest better balance.
Timed Up and Go test (TUG) | 2 minutes
  The TUG test will be used as an index of mobility of the elderly and stroke patients.66 The TUG test measures the time it takes a participant to rise from a chair, walk 3 m, and then return to the chair and sit down. The TUG test will be administered under the single-task and dual-task conditions. In dual-task condition, participants will be asked to perform the TUG test while carrying a tray with glasses (dual-TUG). The instruction for dual-TUG test is to walk with your comfortable speed and carry this tray in front of you with both hands without dropping glasses on the tray.
Activity-specific balance confidence scale (ABC) | 3 minutes
  The ABC will be used to determine self-reported confidence when performing 16 different daily activities, such as walking around the house, walking up and down stairs, and walking on slippery floors. A confidence rating scale ranges from 0% to 100%, with 0% indicating no confidence, and 100% indicating full confidence.
Fugl-Meyer Assessment (FMA) | 5 minutes
  The FMA motor subscale will be used to measure voluntary lower limb motor function in stroke participants with a 3-point ordinal scale on each item (0-cannot perform, 1-performs partially, 2-performs fully) (maximum: 34).
Functional Independent Measurement (FIM) | 5 minutes
  The FIM will be used to assess daily function. The level of participants' disability indicates the burden of caring for them and items are scored on the basis of how much assistance is required for participants to carry out activities of daily living. The FIM consists of 18 items grouped into 6 subscales: self-care, sphincter control, transfer, locomotion, communication, and social cognition ability. Each item is rated from 1 to 7 (max. score 126) based on the required level of assistance to perform the tasks.
Nottingham Extended Activities of Daily Living Scale (NEADL) | 5 minutes
  The NEADL was developed to assess the level of independence in instrumental activity of daily living of stroke patients after hospital discharge. It has four subscales (mobility, domestic, leisure and kitchen) and consists of 22 items scored on the basis of the requirement for help in performing the activity described. The subjects will be asked what they actually did but not what they could do to assess their real daily performance and their level of independence in daily life rather than their capabilities. Items will be scored from 0 to 3 points and summed to provide an overall score, with higher scores indicative of better activities participation.
Stroke Impact Scale Version 3.0 (SIS 3.0) | 10 minutes
  Health-related quality of life will be measured using the SIS 3.0, which is specific to the stroke population. The SIS 3.0 contains 59 items measuring 8 domains (i.e., strength, hand function, Activities of Daily Living/Instrumental Activities of Daily Living [ADL/IADL], mobility, communication, emotion. memory and thinking and participation) with a single item assessing perceived overall recovery from stroke. Items are rated on a 5-point Likert scale with lower scores indicating greater difficulty in task completion during the past week. Aggregate scores, ranges from 0 to 100, are generated for each domain.
Fall rate | 2 minutes
  Participants will be followed prospectively over a period of three months using a falls diary to document their falls event. To assure higher accuracy, participants will also receive monthly follow-up telephone calls to remind them to update their falls diary and the number of falls participants has been fallen in the previous month will be recorded. Participants will be categorized as multiple fallers (≧2 falls), single fallers (1 falls), and non-fallers (no falls) according to information from the falls diaries and monthly follow-up telephone calls.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ling Chuang, Chuang, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chuang LL, Hsu AL, Lin YH, Yu MH, Hu GC, Ou YC, Wong AM. Multimodal training with dual-task enhances immediate and retained effects on dual-task effects of gait speed not by cognitive-motor trade-offs in stroke survivors: a randomized controlled trial. Disabil Rehabil. 2025 Mar;47(5):1194-1203. doi: 10.1080/09638288.2024.2365986. Epub 2024 Jun 17. PMID 38885066